CLINICAL TRIAL: NCT00531752
Title: A Phase Iia, Randomized, Double Blind, Placebo Controlled, Three-treatment, Two-period Crossover Study Of The Efficacy And Safety Of Two Doses Of Pf-03654746 In Adults With Attention Deficit Hyperactivity Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of Two Doses of PF-03654746 in Adults With Attention Deficit Hyperactivity Disorder (ADHD).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A8801004; 3-WK, CO MTD IN ADULTS W/ADHD (Other: Alias Study Number)
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — N-ethyl-3-fluoro-3-(3-fluoro-4-(pyrrolidinylmethyl)phenyl)cyclobutanecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Flexible Dose (Experimental)
  Interventions: Drug: PF-03654746
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo capsules
- Fixed Dose (Experimental)
  Interventions: Drug: PF-03654746

INTERVENTIONS:
Drug: PF-03654746 — Dosage Form: 0.5 mg capsules of PF-03654746 Dosage: 0.5 mg QD for Days 1-7, then 1.0 mg QD Days 8-14, then 2.0 mg QD Days 15-21
  Arms: Flexible Dose
Drug: Placebo capsules — Dosage Form: matching placebo capsules Dosage: Subjects will take two placebo capsules each morning throughout the 3 week double-blind treatment placebo treatment period.
  Arms: Placebo
Drug: PF-03654746 — Dosage Form: 0.5 mg capsules of PF-03654746 Dosage: 1 mg (2 x 0.5 mg capsules) of PF-03654746 given daily for three weeks
  Arms: Fixed Dose

SUMMARY:
The purpose of this study is to determine whether PF-03654746 is effective in the treatment of Adult Attention Deficit Hyperactivity Disorder (ADHD). This will be a randomized, double-blind, crossover study in which adults with ADHD will receive 3 weeks of treatment with PF-03654746, either a low dose (1 mg), or flexible dose (0.50 mg titrated up to 2 mg), and 3 weeks of placebo. A washout period will separate the 2 treatment periods. Participants will be required to washout of prior ADHD medication before entering the study. Participants will be required to come to the site for 10 visits over approximately a 10-week period.

ELIGIBILITY:
Inclusion Criteria:

Subjects with a diagnosis of Attention Deficit Hyperactivity Disorder, based on clinical assessment and interview.

Male and female outpatients. Subjects with a diagnosis of Attention Deficit Hyperactivity Disorder, based on clinical assessment and interview.

Female subjects must be of non-childbearing potential.

Exclusion Criteria:

Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular (including hypertension), hepatic, neurologic, or allergic disease.

Current or lifetime history of psychosis or bipolar disorder; any current anxiety disorder (with the exception of social or specific phobia), or substance abuse or dependence in the past 6 months.

Current episode of Major Depression or episode within the last 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Bay Area Research Institute, Lafayette, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - The University of Illinois at Chicago, Institute for Juvenile Research, Chicago, Illinois
  - Massachusetts General Hospital, ADHD Program, Cambridge, Massachusetts
  - New York University School of Medicine, New York, New York
  - NeuroScience, Inc, Herndon, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8801004&StudyName=A%20Study%20to%20Evaluate%20the%20Efficacy%20and%20Safety%20of%20Two%20Doses%20of%20PF-03654746%20in%20Adults%20with%20Attention%20Deficit%20Hyperactivity%20Disorder%20%28ADH

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First, Then PF-03654746 (Low Dose): Placebo matched to PF-03654746 capsule orally once daily for 3 weeks in first double-blind (DB) intervention period and then low dose of PF-03654746 capsule 1 milligram (mg) orally once daily for 3 weeks in second DB intervention period. A washout period of at least 7 days was maintained between each treatment period.
- PF-03654746 (Low Dose) First, Then Placebo: Low dose of PF-03654746 capsule 1 mg orally once daily for 3 weeks in first DB intervention period and then placebo matched to PF-03654746 capsule orally once daily for 3 weeks in second DB intervention period. A washout period of at least 7 days was maintained between each treatment period.
- Placebo First, Then PF-03654746 (Flexible Dose): Placebo matched to PF-03654746 capsule orally once daily in the first DB intervention period and then PF-03654746 capsule 0.5 mg orally once daily in the first week, PF-03654746 capsule 1 mg orally once daily in the second week and PF-03654746 2 mg orally once daily in the third week, depending upon the investigator's discretion and tolerability, in the second DB intervention period. A washout period of at least 7 days was maintained between each treatment period.
- PF-03654746 (Flexible Dose) First, Then Placebo: PF-03654746 capsule 0.5 mg orally once daily in the first week, PF-03654746 capsule 1 mg orally once daily in the second week and PF-03654746 2 mg orally once daily in the third week, depending upon the investigator's discretion and tolerability, in the first DB intervention period and then placebo matched to PF-03654746 capsule orally once daily in the second DB intervention period. A washout period of at least 7 days was maintained between each treatment period.
Period: First Double-blind Intervention Period
Arm/Group | Placebo First, Then PF-03654746 (Low Dose) | PF-03654746 (Low Dose) First, Then Placebo | Placebo First, Then PF-03654746 (Flexible Dose) | PF-03654746 (Flexible Dose) First, Then Placebo
Started | 17 | 17 | 16 | 16
Treated | 16 | 17 | 16 | 16
Completed | 11 | 13 | 9 | 13
Not Completed | 6 | 4 | 7 | 3
Not completed — Adverse Event | 2 | 0 | 1 | 1
Not completed — Other | 1 | 4 | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Randomized but not treated | 1 | 0 | 0 | 0
Period: Wash-out Period (at Least 7 Days)
Arm/Group | Placebo First, Then PF-03654746 (Low Dose) | PF-03654746 (Low Dose) First, Then Placebo | Placebo First, Then PF-03654746 (Flexible Dose) | PF-03654746 (Flexible Dose) First, Then Placebo
Started | 11 | 13 | 9 | 13
Completed | 11 | 13 | 9 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Second Double-blind Intervention Period
Arm/Group | Placebo First, Then PF-03654746 (Low Dose) | PF-03654746 (Low Dose) First, Then Placebo | Placebo First, Then PF-03654746 (Flexible Dose) | PF-03654746 (Flexible Dose) First, Then Placebo
Started | 11 | 13 | 9 | 13
Completed | 9 | 11 | 9 | 11
Not Completed | 2 | 2 | 0 | 2
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First, Then PF-03654746 (Low Dose) | PF-03654746 (Low Dose) First, Then Placebo | Placebo First, Then PF-03654746 (Flexible Dose) | PF-03654746 (Flexible Dose) First, Then Placebo | Total
Number analyzed (Participants) | 16 | 17 | 16 | 16 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (12.6) | 38.4 (10.6) | 37.9 (10.2) | 35.9 (9.6) | 37.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 16 | 17 | 16 | 16 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Adult Attention Deficit Hyperactivity Disorder (ADHD) Investigator Symptom Rating Scale (AISRS) Total Score at Week 3
Description: AISRS: an 18-item scale administered by the investigator. It included 9 items that evaluated symptoms of inattention and 9 items that evaluated symptoms of impulsivity and hyperactivity. Each item was rated from 0 (none) to 3 (severe). AISRS total score was calculated as sum of all the items on the scale and ranged from 0 to 54. A higher score corresponded to a worse severity of ADHD.
Time Frame: Baseline, Week 3
Population: Per Protocol (PP) set: all participants included in full analysis set (FAS=who received at least[>=]1 dose of randomized study drug,had baseline and >=1 post-baseline measurement of primary efficacy variable)and had no major protocol violation affecting primary efficacy variable. n=participants evaluable at specified time points for each arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PF-03654746 (Low Dose): PF-03654746 capsule 1 mg orally once daily for 3 weeks in first or second DB intervention period.
- PF-03654746 (Flexible Dose): PF-03654746 capsule 0.5 mg orally once daily in the first week, PF-03654746 capsule 1 mg orally once daily in the second week and PF-03654746 2 mg orally once daily in the third week, depending upon the investigator's discretion and tolerability, in first or second DB intervention period.
- Placebo: Placebo matched to PF-03654746 orally once daily for 3 weeks in first or second DB intervention period.
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 27 | 22 | 52
units on a scale
  Baseline (n=27, 22, 52) | 36.778 (8.5545) | 38.273 (4.8715) | 36.135 (7.3592)
  Change at Week 3 (n=25, 21, 48) | -7.196 (8.7318) | -5.745 (9.9824) | -6.789 (8.5734)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.6749, Mixed Models Analysis — P-values are not adjusted for multiple comparisons; Least Squares (LS) Mean Difference = 0.7947, 80% CI 2-sided [-1.649 to 3.2383], Standard Error of Mean 1.8848 — Positive value for the LS mean difference indicates the estimate favors placebo
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4886, Mixed Models Analysis — P-values are not adjusted for multiple comparisons; LS Mean Difference = 1.4176, 80% CI 2-sided [-1.218 to 4.0533], Standard Error of Mean 2.0343 — Positive value for the LS mean difference indicates the estimate favors placebo

2. Secondary Outcome: Change From Baseline in Adult Attention Deficit Hyperactivity Disorder (ADHD) Investigator Symptom Rating Scale (AISRS) Total Score at Week 1 and 2
Description: as for outcome 1
Time Frame: Baseline, Week 1, 2
Population: PP analysis set:all participants included in FAS and had no major protocol violation affecting primary efficacy variable. Here 'N' (number of participants analyzed) signifies participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 26 | 22 | 50
units on a scale
  Week 1 (n=26, 22, 50) | -4.942 (6.2005) | -3.591 (8.3476) | -5.524 (7.4545)
  Week 2 (n=23, 20, 46) | -6.022 (7.1486) | -5.7 (7.8143) | -7.109 (6.6139)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 1: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.5643, Mixed Models Analysis; LS Mean Difference = 1.0250, 80% CI 2-sided [-1.262 to 3.3121], Standard Error of Mean 1.7713
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3107, Mixed Models Analysis; LS Mean Difference = 1.9146, 80% CI 2-sided [-0.5100 to 4.3392], Standard Error of Mean 1.8777
Statistical Analysis 3: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 2: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.1196, Mixed Models Analysis; LS Mean Difference = 2.3154, 80% CI 2-sided [0.41601 to 4.2148], Standard Error of Mean 1.4638
Statistical Analysis 4: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.3872, Mixed Models Analysis; LS Mean Difference = 1.3288, 80% CI 2-sided [-0.6490 to 3.3065], Standard Error of Mean 1.5240

3. Secondary Outcome: Percentage of Participants With at Least 30 Percent Decrease From Baseline in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score
Description: as for outcome 1
Time Frame: Week 1, 2, 3
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 26 | 22 | 50
percentage of participants
  Week 1 (n=26, 22, 50) | 15.385 | 13.636 | 24
  Week 2 (n=23, 20, 46) | 26.087 | 30 | 30.435
  Week 3 (n=25, 21, 48) | 24 | 23.81 | 29.167

4. Secondary Outcome: Percentage of Participants With 1 or 2 Score on Clinical Global Impression-Severity Scale (CGI-S)
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected. Participants with a score of 1 (normal - not ill at all) or 2 (borderline mentally ill) are reported.
Time Frame: Week 1, 2, 3
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 26 | 22 | 50
percentage of participants
  Week 1 (n=26, 22, 50) | 3.846 | 4.545 | 2
  Week 2 (n=23, 20, 49) | 0.0 | 5 | 4.082
  Week 3 (n=25, 21, 50) | 8 | 4.762 | 6

5. Secondary Outcome: Percentage of Participants With Less Than or Equal to 18 Score on Adult ADHD Investigator Symptom Rating Scale (AISRS)
Description: as for outcome 1
Time Frame: Week 1, 2, 3
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 26 | 22 | 50
percentage of participants
  Week 1 (n=26, 22, 50) | 11.538 | 4.545 | 14
  Week 2 (n=23, 20, 46) | 21.739 | 10 | 13.043
  Week 3 (n=25, 21, 48) | 16 | 14.286 | 16.667

6. Secondary Outcome: Percentage of Participants With Sustained Response of at Least 30 Percent Decrease From Baseline in Time-Sensitive ADHD Symptom Scale (TASS) Total Score
Description: TASS: a time sensitive 18-item questionnaire completed by the participant that measured the severity of current ADHD symptoms. It included 9 items that evaluate symptoms of inattention sub-scale and 9 items that evaluate symptoms of impulsivity and hyperactivity sub-scale. Each item was rated from 0 (none) to 3 (severe). TASS total score was calculated as sum of all the items on the scale and ranged from 0 to 54. A higher total score corresponds to a worse severity of ADHD. TASS was administered each day from Day 1 to 14 and on Day 21 in each intervention period. Participants with sustained response were those who had at least 30 percent decrease from baseline in TASS total score, which was maintained at all visits up to the time of assessment. Sustained responders at Day 7, 14 and 21 were analyzed.
Time Frame: Day 7, 14, 21
Population: PP analysis set: all participants included in FAS and had no major protocol violation affecting primary efficacy variable. Here 'N' (number of participants analyzed) signifies participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 21 | 18 | 45
percentage of participants
  Day 7 (n=21, 18, 45) | 38.095 | 27.778 | 33.333
  Day 14 (n=17, 16, 35) | 23.529 | 31.25 | 31.429
  Day 21 (n=9, 6, 22) | 33.333 | 16.667 | 40.909

7. Secondary Outcome: Change From Baseline in Adult ADHD Investigator Symptom Rating Scale (AISRS) Subscale Scores at Week 1, 2 and 3
Description: AISRS: an 18-item scale administered by the investigator. It included 9 items that evaluated symptoms of inattention and 9 items that evaluated symptoms of impulsivity and hyperactivity. Each item was rated from 0 (none) to 3 (severe). The AISRS inattention and hyperactive/impulsive total subscale score range from 0 to 27. A higher total subscale score corresponded to a worse severity of ADHD inattention or hyperactivity/impulsivity.
Time Frame: Baseline, Week 1, 2, 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 26 | 22 | 50
units on a scale
  Week 1: Inattention (n=26, 22, 50) | -3.423 (3.6241) | -1.636 (4.7338) | -3.36 (4.3986)
  Week 2: Inattention (n=23, 20, 46) | -4.326 (5.2627) | -2.65 (4.5541) | -4.022 (4.2985)
  Week 3: Inattention (n=25, 21, 48) | -4.085 (5.7909) | -3.31 (5.8019) | -3.719 (5.195)
  Week 1: Hyperactivity/Impulsivity (n=26, 22, 50) | -1.519 (3.708) | -1.955 (4.0027) | -2.164 (3.7001)
  Week 2: Hyperactivity/Impulsivity (n=23, 20, 46) | -1.696 (3.1935) | -3.05 (3.9766) | -3.087 (3.2614)
  Week 3: Hyperactivity/Impulsivity (n=25, 21, 48) | -3.111 (4.1894) | -2.435 (4.8666) | -3.07 (4.2411)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 1 (Inattention): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.8708, Mixed Models Analysis; LS Mean Difference = 0.1677, 80% CI 2-sided [-1.162 to 1.4971], Standard Error of Mean 1.0269
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0927, Mixed Models Analysis; LS Mean Difference = 1.8607, 80% CI 2-sided [0.44874 to 3.2726], Standard Error of Mean 1.0912
Statistical Analysis 3: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 1 (Hyperactivity/Impulsivity): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.3405, Mixed Models Analysis; LS Mean Difference = 0.8660, 80% CI 2-sided [-0.3008 to 2.0329], Standard Error of Mean 0.9037
Statistical Analysis 4: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 7, analysis 3]; Test type: Superiority or Other; p = 0.8665, Mixed Models Analysis; LS Mean Difference = 0.1623, 80% CI 2-sided [-1.080 to 1.4047], Standard Error of Mean 0.9622
Statistical Analysis 5: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 2 (Inattention): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.6901, Mixed Models Analysis; LS Mean Difference = 0.3886, 80% CI 2-sided [-0.8694 to 1.6466], Standard Error of Mean 0.9694
Statistical Analysis 6: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; p = 0.1790, Mixed Models Analysis; LS Mean Difference = 1.3779, 80% CI 2-sided [0.06498 to 2.6908], Standard Error of Mean 1.0114
Statistical Analysis 7: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 2 (Hyperactivity/Impulsivity): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0156, Mixed Models Analysis; LS Mean Difference = 1.8759, 80% CI 2-sided [0.90156 to 2.8502], Standard Error of Mean 0.7508
Statistical Analysis 8: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; p = 0.9573, Mixed Models Analysis; LS Mean Difference = -0.04217, 80% CI 2-sided [-1.060 to 0.97559], Standard Error of Mean 0.7842
Statistical Analysis 9: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Inattention): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.8986, Mixed Models Analysis; LS Mean Difference = 0.1602, 80% CI 2-sided [-1.462 to 1.7820], Standard Error of Mean 1.2517
Statistical Analysis 10: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 7, analysis 9]; Test type: Superiority or Other; p = 0.6204, Mixed Models Analysis; LS Mean Difference = 0.6688, 80% CI 2-sided [-1.071 to 2.4086], Standard Error of Mean 1.3437
Statistical Analysis 11: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Hyperactivity/Impulsivity): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.5759, Mixed Models Analysis; LS Mean Difference = 0.4920, 80% CI 2-sided [-0.6421 to 1.6261], Standard Error of Mean 0.8742
Statistical Analysis 12: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 7, analysis 11]; Test type: Superiority or Other; p = 0.3603, Mixed Models Analysis; LS Mean Difference = 0.8750, 80% CI 2-sided [-0.3552 to 2.1051], Standard Error of Mean 0.9488

8. Secondary Outcome: Change From Baseline in Time-Sensitive ADHD Symptom Scale (TASS) Total Score on Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 21
Description: TASS: a time sensitive 18-item questionnaire completed by the participant that measured the severity of current ADHD symptoms. It included 9 items that evaluate symptoms of inattention sub-scale and 9 items that evaluate symptoms of impulsivity and hyperactivity sub-scale. Each item was rated from 0 (none) to 3 (severe). TASS total score was calculated as sum of all the items on the scale and ranged from 0 to 54. A higher total score corresponded to a worse severity of ADHD. TASS was administered each day from Day 1 to 14 and on Day 21 in each intervention period.
Time Frame: Baseline, Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 21
Population: Analysis population included all participants in PP analysis set and 1 additional participant in PF-03654746 (Flexible Dose) for whom the post-baseline data was available.'N' (number of participants analyzed)=evaluable participants for this measure and 'n'= evaluable participants for this measure at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 27 | 23 | 50
units on a scale
  Day 1 (n=25, 22, 50) | -0.46 (5.3384) | 2.205 (14.9217) | -4.75 (6.7221)
  Day 2 (n=25, 21, 49) | -1.78 (6.8679) | -0.952 (13.4433) | -6.031 (10.2938)
  Day 3 (n=26, 21, 49) | -2.798 (12.1305) | -3.857 (10.0476) | -3.51 (10.3282)
  Day 4 (n=26, 22, 46) | -4.981 (8.8346) | -1.068 (14.4018) | -3.761 (9.682)
  Day 5 (n=26, 23, 49) | -4.942 (7.7153) | -1.87 (10.2239) | -6.622 (8.9353)
  Day 6 (n=27, 22, 44) | -5.833 (7.3183) | -3.205 (10.5984) | -6.841 (9.9573)
  Day 7 (n=21, 18, 45) | -6.381 (7.7619) | -6.222 (11.2736) | -4.789 (9.7044)
  Day 8 (n=21, 19, 46) | -5.952 (7.0709) | -6.526 (9.7389) | -5.272 (9.804)
  Day 9 (n=21, 18, 45) | -4.238 (6.1352) | -5.889 (9.9979) | -5.889 (10.8664)
  Day 10 (n=20, 20, 46) | -5.75 (6.9689) | -7.525 (9.6579) | -6.837 (10.7755)
  Day 11 (n=21, 20, 46) | -5.619 (6.7341) | -5.875 (11.2377) | -6.924 (10.4371)
  Day 12 (n=20, 18, 44) | -6.45 (7.3947) | -6.167 (10.3099) | -6.295 (10.3622)
  Day 13 (n=22, 19, 43) | -6.091 (6.4284) | -5.658 (11.024) | -7.488 (7.9279)
  Day 14 (n=17, 16, 35) | -5.147 (6.7818) | -7.5 (11.0559) | -2.506 (25.19)
  Day 21 (n=9, 6, 22) | -9.889 (7.474) | -4.583 (8.4346) | -8.295 (8.299)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 1: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0392, Mixed Models Analysis; LS Mean Difference = 3.5306, 80% CI 2-sided [1.3659 to 5.6952], Standard Error of Mean 1.6664
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; LS Mean Difference = 6.9344, 80% CI 2-sided [4.6177 to 9.2512], Standard Error of Mean 1.7848
Statistical Analysis 3: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 2: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0547, Mixed Models Analysis; LS Mean Difference = 4.2888, 80% CI 2-sided [1.4544 to 7.1232], Standard Error of Mean 2.1861
Statistical Analysis 4: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; p = 0.0176, Mixed Models Analysis; LS Mean Difference = 5.6799, 80% CI 2-sided [2.6655 to 8.6943], Standard Error of Mean 2.3261
Statistical Analysis 5: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 3: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.7750, Mixed Models Analysis; LS Mean Difference = 0.7203, 80% CI 2-sided [-2.530 to 3.9704], Standard Error of Mean 2.5085
Statistical Analysis 6: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority or Other; p = 0.9874, Mixed Models Analysis; LS Mean Difference = -0.04276, 80% CI 2-sided [-3.521 to 3.4357], Standard Error of Mean 2.6874
Statistical Analysis 7: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 4: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.7799, Mixed Models Analysis; LS Mean Difference = -0.6252, 80% CI 2-sided [-3.513 to 2.2629], Standard Error of Mean 2.2268
Statistical Analysis 8: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.1881, Mixed Models Analysis; LS Mean Difference = 3.1136, 80% CI 2-sided [0.08338 to 6.1438], Standard Error of Mean 2.3365
Statistical Analysis 9: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 5: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.4032, Mixed Models Analysis; LS Mean Difference = 1.6575, 80% CI 2-sided [-0.8944 to 4.2094], Standard Error of Mean 1.9677
Statistical Analysis 10: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 9]; Test type: Superiority or Other; p = 0.0059, Mixed Models Analysis; LS Mean Difference = 5.9254, 80% CI 2-sided [3.2314 to 8.6193], Standard Error of Mean 2.0796
Statistical Analysis 11: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 6: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.6067, Mixed Models Analysis; LS Mean Difference = 1.0921, 80% CI 2-sided [-1.643 to 3.8273], Standard Error of Mean 2.1098
Statistical Analysis 12: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 11]; Test type: Superiority or Other; p = 0.0614, Mixed Models Analysis; LS Mean Difference = 4.2785, 80% CI 2-sided [1.3709 to 7.1860], Standard Error of Mean 2.2424
Statistical Analysis 13: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 7: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.7476, Mixed Models Analysis; LS Mean Difference = -0.7149, 80% CI 2-sided [-3.584 to 2.1546], Standard Error of Mean 2.2086
Statistical Analysis 14: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.5863, Mixed Models Analysis; LS Mean Difference = -1.3355, 80% CI 2-sided [-4.499 to 1.8284], Standard Error of Mean 2.4396
Statistical Analysis 15: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 8: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.9591, Mixed Models Analysis; LS Mean Difference = -0.1058, 80% CI 2-sided [-2.771 to 2.5593], Standard Error of Mean 2.0529
Statistical Analysis 16: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 15]; Test type: Superiority or Other; p = 0.8442, Mixed Models Analysis; LS Mean Difference = -0.4352, 80% CI 2-sided [-3.294 to 2.4238], Standard Error of Mean 2.2048
Statistical Analysis 17: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 9: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.1977, Mixed Models Analysis; LS Mean Difference = 2.6876, 80% CI 2-sided [0.01391 to 5.3613], Standard Error of Mean 2.0533
Statistical Analysis 18: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 17]; Test type: Superiority or Other; p = 0.4235, Mixed Models Analysis; LS Mean Difference = 1.8149, 80% CI 2-sided [-1.108 to 4.7375], Standard Error of Mean 2.2467
Statistical Analysis 19: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 10: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.1882, Mixed Models Analysis; LS Mean Difference = 2.6424, 80% CI 2-sided [0.07015 to 5.2147], Standard Error of Mean 1.9753
Statistical Analysis 20: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p = 0.5555, Mixed Models Analysis; LS Mean Difference = 1.2105, 80% CI 2-sided [-1.440 to 3.8615], Standard Error of Mean 2.0376
Statistical Analysis 21: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 11: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.1533, Mixed Models Analysis; LS Mean Difference = 3.1804, 80% CI 2-sided [0.33169 to 6.0292], Standard Error of Mean 2.1934
Statistical Analysis 22: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 21]; Test type: Superiority or Other; p = 0.3697, Mixed Models Analysis; LS Mean Difference = 2.0511, 80% CI 2-sided [-0.8912 to 4.9934], Standard Error of Mean 2.2662
Statistical Analysis 23: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 12: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.4652, Mixed Models Analysis; LS Mean Difference = 1.7640, 80% CI 2-sided [-1.352 to 4.8801], Standard Error of Mean 2.3939
Statistical Analysis 24: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 23]; Test type: Superiority or Other; p = 0.8626, Mixed Models Analysis; LS Mean Difference = 0.4377, 80% CI 2-sided [-2.830 to 3.7058], Standard Error of Mean 2.5148
Statistical Analysis 25: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 13: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0261, Mixed Models Analysis; LS Mean Difference = 3.7114, 80% CI 2-sided [1.6105 to 5.8122], Standard Error of Mean 1.6168
Statistical Analysis 26: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p = 0.1895, Mixed Models Analysis; LS Mean Difference = 2.2644, 80% CI 2-sided [0.05330 to 4.4756], Standard Error of Mean 1.7026
Statistical Analysis 27: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 14: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.4994, Mixed Models Analysis; LS Mean Difference = 2.1151, 80% CI 2-sided [-1.961 to 6.1913], Standard Error of Mean 3.0732
Statistical Analysis 28: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 27]; Test type: Superiority or Other; p = 0.2945, Mixed Models Analysis; LS Mean Difference = 3.5616, 80% CI 2-sided [-0.8226 to 7.9458], Standard Error of Mean 3.3113
Statistical Analysis 29: Comparison: PF-03654746 (Low Dose) vs Placebo; Day 21: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.8056, Mixed Models Analysis; LS Mean Difference = -0.7306, 80% CI 2-sided [-4.622 to 3.1613], Standard Error of Mean 2.9257
Statistical Analysis 30: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 29]; Test type: Superiority or Other; p = 0.3922, Mixed Models Analysis; LS Mean Difference = 3.3672, 80% CI 2-sided [-1.725 to 8.4592], Standard Error of Mean 3.8657

9. Secondary Outcome: Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score at Week 3
Description: The MADRS scale measures the depression level of a participant. It is administered as a semi-structured clinician interview. The total score is derived by adding the scores of the following 10 items: (1) Apparent sadness; (2) Reported sadness; (3) Inner tension; (4) Reduced sleep; (5) Reduced appetite; (6) Concentration difficulties; (7) Lassitude; (8) Inability to feel; (9) Pessimistic thoughts; (10) Suicidal thoughts. Each item is scored using a 6-point scale which ranges from 0 to 6 (a higher score indicates increased severity). The total score range was 0 to 60 where 0 indicates no depression and 60 indicates severely depressed.
Time Frame: Baseline, Week 3
Population: PP analysis set: all participants included in FAS and had no major protocol violation affecting primary efficacy variable. Here 'n' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 27 | 22 | 52
units on a scale
  Baseline (n=27, 22, 52) | 6.63 (3.9918) | 7.773 (5.0231) | 6.962 (4.5631)
  Change at Week 3 (n=21, 19, 42) | -2.19 (3.9353) | -1.289 (3.728) | -0.524 (5.1572)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3: Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0913, Mixed Models Analysis; LS Mean Difference = -1.5069, 80% CI 2-sided [-2.643 to -0.3705], Standard Error of Mean 0.8744
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority or Other; p = 0.8216, Mixed Models Analysis; LS Mean Difference = -0.2078, 80% CI 2-sided [-1.399 to 0.98326], Standard Error of Mean 0.9165

10. Secondary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) Total Score at Week 3
Description: HAM-A is a clinician-rated 14 item scale that provides an overall measure of global anxiety, including psychic (mental agitation and psychological distress) and somatic (physical complaints related to anxiety) symptoms. Each item was scored on a scale ranging from 0 (not present) to 4 (very severe) with a total score range of 0 to 56, where higher score indicates greater anxiety.
Time Frame: Baseline, Week 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 27 | 22 | 52
units on a scale
  Baseline (n=27, 22, 52) | 5.333 (3.9223) | 6.045 (3.848) | 5.327 (3.3238)
  Change at Week 3 (n=18, 21, 39) | -0.944 (2.514) | -0.19 (2.5518) | -0.487 (2.7732)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.5466, Mixed Models Analysis; LS Mean Difference = -0.4181, 80% CI 2-sided [-1.313 to 0.47668], Standard Error of Mean 0.6887
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.9705, Mixed Models Analysis; LS Mean Difference = -0.02518, 80% CI 2-sided [-0.9035 to 0.85312], Standard Error of Mean 0.6772

11. Secondary Outcome: Change From Baseline in ADHD Impact Module - Adults (AIM-A) Subscale Score at Week 3
Description: AIM-A: 66 item questionnaire completed by the participant to assess the impact of ADHD on the participant's quality of life. It is comprised of 4 global quality of life (QoL) items (current quality of life item [CQoLI], range:1 to 10; global limitation item [GLI]: range:1 to 4, on the right track item [RTI], range:1 to 3, more good days [GD] than bad days [BD], range:1 to 5, higher scores indicate a better QoL for all the 4 QoL items) and 6 multi-item subscales (living with ADHD, general well-being, performance and daily functioning [PDF], relationships and communication [R/C], Impact of symptoms-bother/concern [IS-B/C] scale, and impact of symptoms-interference [IS-I] scale). Participants responded to each item of multi-item subscale using a likert scale ranging from 1 (strongly agree) to 5 (strongly disagree). Multi-item subscale scores were calculated as an average of scores for the contributing items and transformed into 0 to 100 score where higher scores indicate a better QoL.
Time Frame: Baseline, Week 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 27 | 22 | 52
units on a scale
  Baseline: CQoLI (n=27, 22, 52) | 6.481 (1.2746) | 6.409 (1.1406) | 6.423 (1.1219)
  Baseline: GLI (n=27, 22, 52) | 1.815 (0.7091) | 1.705 (0.7505) | 1.663 (0.624)
  Baseline: RTI (n=27, 22, 52) | 1.944 (0.5938) | 2.068 (0.3872) | 1.99 (0.4999)
  Baseline: More GD than BD (n=27, 22, 52) | 2.259 (0.7642) | 2.682 (0.8803) | 2.529 (0.8069)
  Baseline: Living with ADHD (n=27, 22, 52) | 53.935 (9.587) | 49.773 (12.4202) | 51.058 (10.5294)
  Baseline: General well-being (n=27, 22, 52) | 54.377 (11.1639) | 50.413 (17.2322) | 50.83 (13.2045)
  Baseline: PDF (n=27, 22, 52) | 37.176 (15.634) | 34.489 (15.3756) | 34.688 (13.5081)
  Baseline: R/C (n=27, 22, 52) | 65.856 (16.2652) | 57.955 (15.7281) | 61.358 (14.7036)
  Baseline: IS-B/C (n=27, 22, 52) | 44.753 (16.8364) | 42.235 (19.7475) | 42.201 (16.7033)
  Baseline: IS-I (n=27, 22, 52) | 47.994 (10.1284) | 46.78 (9.1366) | 46.768 (8.8729)
  Change at Week 3: CQoLI (n=25, 21, 47) | 0.04 (0.9456) | 0.286 (1.2306) | 0.17 (1.3116)
  Change at Week 3: GLI (n=25, 21, 47) | 0.2 (0.4564) | 0.214 (0.7676) | 0.106 (0.6421)
  Change at Week 3: RTI (n=25, 21, 47) | -0.02 (0.5492) | -0.071 (0.6381) | -0.074 (0.5612)
  Change at Week 3: More GD than BD (n=25, 21, 47) | -0.32 (0.6272) | -0.238 (0.9826) | -0.106 (0.9997)
  Change at Week 3: Living with ADHD (n=25, 21, 47) | 2.55 (4.5712) | 1.905 (5.5145) | 3.005 (7.2121)
  Change at Week 3:General well-being (n=25, 21, 47) | 4.909 (7.1999) | 1.299 (8.9642) | 4.884 (10.3145)
  Change at Week 3: PDF (n=25, 21, 47) | 12.65 (14.0698) | 11.488 (21.7501) | 10.718 (18.3226)
  Change at Week 3: R/C (n=25, 21, 47) | 5.125 (13.0457) | 0.298 (16.3773) | 3.358 (13.4687)
  Change at Week 3: IS-B/C (n=25, 21, 47) | 3 (12.9465) | 0.463 (18.6097) | 7.417 (13.7471)
  Change at Week 3: IS-I (n=25, 21, 47) | 2.389 (8.2023) | 0.463 (9.3204) | 2.896 (10.6124)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (CQoL): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.7415, Mixed Models Analysis; LS Mean Difference = -0.09953, 80% CI 2-sided [-0.4892 to 0.29012], Standard Error of Mean 0.3001
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.8822, Mixed Models Analysis; LS Mean Difference = 0.04804, 80% CI 2-sided [-0.3703 to 0.46640], Standard Error of Mean 0.3227
Statistical Analysis 3: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (GLI): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.3414, Mixed Models Analysis; LS Mean Difference = 0.1250, 80% CI 2-sided [-0.0439 to 0.29385], Standard Error of Mean 0.1302
Statistical Analysis 4: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 11, analysis 3]; Test type: Superiority or Other; p = 0.4642, Mixed Models Analysis; LS Mean Difference = 0.1044, 80% CI 2-sided [-0.0793 to 0.28814], Standard Error of Mean 0.1418
Statistical Analysis 5: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (RTI): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.5049, Mixed Models Analysis; LS Mean Difference = 0.06109, 80% CI 2-sided [-0.0571 to 0.17926], Standard Error of Mean 0.09093
Statistical Analysis 6: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 11, analysis 5]; Test type: Superiority or Other; p = 0.4332, Mixed Models Analysis; LS Mean Difference = 0.07917, 80% CI 2-sided [-0.0510 to 0.20930], Standard Error of Mean 0.1002
Statistical Analysis 7: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (More GD than BD): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.1678, Mixed Models Analysis; LS Mean Difference = -0.2453, 80% CI 2-sided [-0.4730 to -0.0177], Standard Error of Mean 0.1753
Statistical Analysis 8: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 11, analysis 7]; Test type: Superiority or Other; p = 0.6901, Mixed Models Analysis; LS Mean Difference = 0.07717, 80% CI 2-sided [-0.1726 to 0.32695], Standard Error of Mean 0.1925
Statistical Analysis 9: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Living with ADHD): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.9005, Mixed Models Analysis; LS Mean Difference = 0.1702, 80% CI 2-sided [-1.587 to 1.9274], Standard Error of Mean 1.3540
Statistical Analysis 10: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 11, analysis 9]; Test type: Superiority or Other; p = 0.3330, Mixed Models Analysis; LS Mean Difference = -1.4317, 80% CI 2-sided [-3.333 to 0.46937], Standard Error of Mean 1.4667
Statistical Analysis 11: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (General well-being): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.7551, Mixed Models Analysis; LS Mean Difference = 0.6537, 80% CI 2-sided [-2.051 to 3.3584], Standard Error of Mean 2.0857
Statistical Analysis 12: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.0334, Mixed Models Analysis; LS Mean Difference = -4.8639, 80% CI 2-sided [-7.759 to -1.968], Standard Error of Mean 2.2354
Statistical Analysis 13: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (PDF): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.6519, Mixed Models Analysis; LS Mean Difference = 1.6389, 80% CI 2-sided [-3.050 to 6.3281], Standard Error of Mean 3.6119
Statistical Analysis 14: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 11, analysis 13]; Test type: Superiority or Other; p = 0.7631, Mixed Models Analysis; LS Mean Difference = 1.2007, 80% CI 2-sided [-3.941 to 6.3423], Standard Error of Mean 3.9647
Statistical Analysis 15: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (R/C): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.3034, Mixed Models Analysis; LS Mean Difference = 2.9211, 80% CI 2-sided [-0.7227 to 6.5648], Standard Error of Mean 2.8206
Statistical Analysis 16: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 11, analysis 15]; Test type: Superiority or Other; p = 0.0933, Mixed Models Analysis; LS Mean Difference = -5.0968, 80% CI 2-sided [-8.975 to -1.218], Standard Error of Mean 3.0022
Statistical Analysis 17: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (IS-B/C): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0949, Mixed Models Analysis; LS Mean Difference = -5.0675, 80% CI 2-sided [-8.934 to -1.201], Standard Error of Mean 2.9778
Statistical Analysis 18: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 11, analysis 17]; Test type: Superiority or Other; p = 0.0283, Mixed Models Analysis; LS Mean Difference = -7.3274, 80% CI 2-sided [-11.55 to -3.106], Standard Error of Mean 3.2552
Statistical Analysis 19: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (IS-I): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.1852, Mixed Models Analysis; LS Mean Difference = -2.1505, 80% CI 2-sided [-4.229 to -0.0719], Standard Error of Mean 1.5974
Statistical Analysis 20: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 11, analysis 19]; Test type: Superiority or Other; p = 0.1623, Mixed Models Analysis; LS Mean Difference = -2.5178, 80% CI 2-sided [-4.823 to -0.2127], Standard Error of Mean 1.7732

12. Secondary Outcome: Change From Baseline in Adult ADHD Quality of Life Scale (AAQOL) Subscale Score at Week 3
Description: AAQoL is a 29-item questionnaire consisting of 4 subscales: life productivity (11 items), psychological health ([PH] 6 items), life outlook (7 items) and relationships (5 items). Participants rated each item on a scale ranging from 1 (not at all/never) to 5 (extremely/very often). The scores of each item were then transformed to a 0 to 100 point scale, higher scores indicating better quality of life. The score for each subscale was calculated as the sum of the corresponding item scores. Total score ranges were: life productivity (0 to 1100), psychological health (0 to 600), life outlook (0 to 700) and relationships (0 to 500), where higher subscale score indicates better quality of life for each subscale.
Time Frame: Baseline, Week 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 27 | 22 | 52
units on a scale
  Baseline: Life productivity (n=27, 22, 52) | 306.481 (109.9809) | 292.045 (72.5334) | 281.25 (107.9982)
  Baseline: Psychological health (n=27, 22, 52) | 163.889 (42.9296) | 146.591 (66.0517) | 167.788 (59.4782)
  Baseline: Life outlook (n=27, 22, 52) | 229.63 (65.7929) | 194.318 (69.8348) | 218.269 (59.0188)
  Baseline: Relationships (n=27, 22, 52) | 152.778 (49.1922) | 154.545 (46.0566) | 163.942 (49.856)
  Change at Week 3: Life productivity (n=25, 21, 47) | 3 (84.1068) | 8.333 (112.7312) | 22.606 (85.7606)
  Change at Week 3: PH (n=25, 21, 47) | 0 (50.5181) | 1.786 (57.1847) | 11.436 (63.9415)
  Change at Week 3: Life outlook (n=25, 21, 47) | -13 (56.9951) | 14.286 (68.9526) | -8.511 (42.6776)
  Change at Week 3: Relationships (n=25, 21, 47) | -1.5 (31.9342) | 1.19 (46.2508) | -3.723 (45.662)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Life productivity): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.5241, Mixed Models Analysis; LS Mean Difference = -11.5791, 80% CI 2-sided [-35.02 to 11.860], Standard Error of Mean 18.0449
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.3065, Mixed Models Analysis; LS Mean Difference = -20.3367, 80% CI 2-sided [-45.89 to 5.2183], Standard Error of Mean 19.6995
Statistical Analysis 3: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Psychological health): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.3831, Mixed Models Analysis; LS Mean Difference = -11.7878, 80% CI 2-sided [-29.15 to 5.5793], Standard Error of Mean 13.4438
Statistical Analysis 4: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 12, analysis 3]; Test type: Superiority or Other; p = 0.3657, Mixed Models Analysis; LS Mean Difference = -13.1401, 80% CI 2-sided [-31.80 to 5.5241], Standard Error of Mean 14.4478
Statistical Analysis 5: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Life outlook): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.8188, Mixed Models Analysis; LS Mean Difference = 2.6660, 80% CI 2-sided [-12.36 to 17.690], Standard Error of Mean 11.5818
Statistical Analysis 6: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 12, analysis 5]; Test type: Superiority or Other; p = 0.0566, Mixed Models Analysis; LS Mean Difference = 24.1011, 80% CI 2-sided [8.0305 to 40.172], Standard Error of Mean 12.4050
Statistical Analysis 7: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Relationships): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.9312, Mixed Models Analysis; LS Mean Difference = 0.7559, 80% CI 2-sided [-10.55 to 12.057], Standard Error of Mean 8.7164
Statistical Analysis 8: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p = 0.5194, Mixed Models Analysis; LS Mean Difference = 6.1138, 80% CI 2-sided [-6.108 to 18.336], Standard Error of Mean 9.4361

13. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Subscale Scores at Week 3
Description: SDS was a participant-rated questionnaire assessing the effect of the participant's symptoms on the 3 domains/subscales: work/school, social life/leisure activities, and family/home management. Each domain was rated on visual analog scale ranges from 0 to 10 where 0=not at all impaired and 10=extremely impaired, and total SDS score was calculated as a sum of all the domains with a score range of 0=not at all impaired to 30=extremely impaired. Disability scores were reported for each of the domains/subscales. Higher scores reflect greater impairment.
Time Frame: Baseline, Week 3
Population: PP analysis set: all participants included in FAS and had no major protocol violation affecting primary efficacy variable. Here 'n' signifies those participants who were evaluable for given subscale at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 27 | 22 | 52
units on a scale
  Baseline: Work/school (n=26, 21, 50) | 6.058 (2.2375) | 6.095 (2.0894) | 6.36 (1.977)
  Baseline: Social life (n=27, 22, 52) | 4.593 (2.0383) | 5.227 (2.5153) | 5.01 (2.0757)
  Baseline: Family life/home (n=27, 22, 52) | 5.019 (2.0357) | 5.705 (2.0393) | 5.673 (1.8335)
  Change at Week 3: Work/school (n=24, 18, 45) | -0.813 (1.3089) | -0.222 (2.2572) | -0.411 (1.7526)
  Change at Week 3: Social life (n=25, 21, 47) | -0.8 (1.75) | -0.619 (2.4592) | -0.436 (1.9043)
  Change at Week 3: Family life/home (n=25, 21, 47) | -0.78 (1.5618) | -0.071 (2.2709) | -0.532 (1.6596)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Work/school): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.3320, Mixed Models Analysis; LS Mean Difference = -0.3255, 80% CI 2-sided [-0.7573 to 0.10622], Standard Error of Mean 0.3320
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.2767, Mixed Models Analysis; LS Mean Difference = 0.4255, 80% CI 2-sided [-0.0769 to 0.92804], Standard Error of Mean 0.3871
Statistical Analysis 3: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Social life): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.3675, Mixed Models Analysis; LS Mean Difference = -0.3661, 80% CI 2-sided [-0.8887 to 0.15660], Standard Error of Mean 0.4028
Statistical Analysis 4: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 13, analysis 3]; Test type: Superiority or Other; p = 0.8141, Mixed Models Analysis; LS Mean Difference = -0.1033, 80% CI 2-sided [-0.6700 to 0.46345], Standard Error of Mean 0.4372
Statistical Analysis 5: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Family life/home): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.6186, Mixed Models Analysis; LS Mean Difference = -0.1854, 80% CI 2-sided [-0.6657 to 0.29495], Standard Error of Mean 0.3702
Statistical Analysis 6: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 13, analysis 5]; Test type: Superiority or Other; p = 0.3720, Mixed Models Analysis; LS Mean Difference = 0.3623, 80% CI 2-sided [-0.1597 to 0.88432], Standard Error of Mean 0.4028

14. Other Pre Specified Outcome: Change From Baseline in Medical Outcome Study - Sleep Scale (MOS-SS) Subscale Scores at Week 1, 2 and 3
Description: Participant-rated 12-item questionnaire to assess sleep quality and quantity. The items contribute to each scale and are averaged to create the 7 subscale scores: sleep disturbance, snoring, awaken short of breath (ASoB) or with a headache, somnolence, sleep adequacy, sleep quantity (range 0 to 24) and optimal sleep, and overall sleep problem index (SPI) I (range 0 to 600) and II. Except for sleep quantity and sleep problem index I, scores are transformed (actual raw score minus lowest possible score divided by possible raw score range* 100); total score range: 0 to 100; higher score = greater intensity of attribute. Except for sleep quantity, higher scores=greater impairment. Scales with at least one item answered was used to generate a scale score.
Time Frame: Baseline, Week 1, 2, 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 27 | 22 | 52
units on a scale
  Baseline: Sleep disturbance (n=27, 22, 52) | 27.894 (19.427) | 34.489 (20.6801) | 29.892 (20.4408)
  Baseline: Snoring (n=26, 22, 51) | 43.462 (29.1125) | 44.091 (32.9009) | 40.784 (29.9895)
  Baseline: ASoB (n=27, 22, 52) | 3.333 (8.7706) | 7.727 (17.7098) | 6.154 (14.1635)
  Baseline: Sleep quantity (n=27, 22, 52) | 6.537 (0.95) | 6.705 (0.9594) | 6.673 (1.0379)
  Baseline: Optimal sleep (n=27, 22, 52) | 1.593 (0.4169) | 1.5 (0.4082) | 1.558 (0.416)
  Baseline: Sleep adequacy (n=26, 22, 51) | 40.962 (22.8044) | 41.364 (26.1944) | 39.804 (23.4512)
  Baseline: Somnolence (n=26, 22, 51) | 31.795 (19.6238) | 32.727 (19.5893) | 30.85 (20.2522)
  Baseline: SPI I (n=26, 22, 51) | 201.538 (69.0329) | 214.091 (109.1377) | 210.196 (87.7836)
  Baseline: SPI II (n=27, 22, 52) | 33.251 (12.8016) | 37.519 (18.3575) | 34.848 (15.5578)
  Change at Week 1: Sleep disturbance (n=26, 22, 50) | 18.245 (30.9066) | 4.489 (23.7105) | -8.263 (18.8354)
  Change at Week 1: Snoring (n=25, 21, 48) | -14.8 (19.1746) | -4.286 (17.7684) | -10.417 (14.1359)
  Change at Week 1: ASoB (n=26, 22, 50) | 4.231 (15.7919) | -2.273 (9.2231) | -1.6 (14.3371)
  Change at Week 1: Sleep quantity (n=25, 22, 48) | -0.42 (1.3204) | -0.114 (0.8442) | 0.198 (1.0249)
  Change at Week 1: Optimal sleep (n=26, 22, 50) | 0 (0.4899) | 0 (0.5345) | -0.14 (0.5349)
  Change at Week 1: Sleep Adequacy (n=25, 22, 49) | -1.8 (15.6045) | -6.818 (27.1041) | -0.408 (21.5985)
  Change at Week 1: Somnolence (n=25, 22, 49) | -8.267 (21.7545) | -1.818 (13.8674) | -1.769 (16.4444)
  Change at Week 1: SPI I (n=25, 22, 49) | 35.2 (81.7068) | 25 (105.9088) | -21.224 (85.9901)
  Change at Week 1: SPI II (n=26, 22, 50) | 7.65 (16.0588) | 2.936 (17.1929) | -3.875 (14.2472)
  Change at Week 2: Sleep disturbance (n=23, 20, 46) | 3.904 (18.0117) | 0.438 (27.3712) | -11.984 (15.9101)
  Change at Week 2: Snoring (n=22, 19, 45) | -12.273 (17.1636) | -17.368 (14.4692) | -12 (14.554)
  Change at Week 2: ASoB (n=23, 20, 46) | 0.435 (11.0693) | 1.5 (14.2441) | -3.478 (11.1987)
  Change at Week 2: Sleep quantity (22, 20, 46) | -0.182 (0.958) | 0.025 (0.8955) | 0.152 (0.9121)
  Change at Week 2: Optimal sleep (n=23, 20, 49) | 0.065 (0.4074) | -0.1 (0.4472) | -0.122 (0.4845)
  Change at Week 2: Sleep Adequacy (n=22, 20, 45) | 7.955 (17.6378) | 4.5 (23.6699) | 6.111 (24.0711)
  Change at Week 2: Somnolence (n=22, 20, 45) | -6.061 (16.9542) | -4.333 (14.3515) | -5.333 (14.6059)
  Change at Week 2: SPI I (n=22, 20, 45) | -15.455 (71.6956) | 1.5 (103.937) | -45.333 (74.8817)
  Change at Week 2: SPI II (n=23, 20, 46) | -0.242 (11.7718) | -1.438 (17.3576) | -8.155 (12.6707)
  Change at Week 3: Sleep disturbance (n=25, 21, 47) | -0.875 (18.0287) | 6.31 (24.7652) | -12.114 (15.1541)
  Change at Week 3: Snoring (n=24, 20, 44) | -7.917 (14.44) | -5.5 (20.1246) | -6.364 (13.6554)
  Change at Week 3: ASoB (n=25, 21, 47) | -0.4 (12.0692) | 6.19 (19.3588) | 1.702 (22.4886)
  Change at Week 3: Sleep quantity (n=24, 20, 47) | -0.354 (0.8658) | -0.025 (0.9244) | 0.16 (1.0638)
  Change at Week 3: Optimal sleep (n=25, 21, 50) | 0.08 (0.4491) | 0 (0.5477) | -0.12 (0.5206)
  Change at Week 3: Sleep Adequacy (n=24, 21, 45) | 3.958 (19.1663) | -2.381 (25.5254) | 3 (17.235)
  Change at Week 3: Somnolence (n=24, 21, 45) | -8.889 (19.5274) | 0.635 (13.3591) | -1.704 (12.4848)
  Change at Week 3: SPI I (n=24, 21, 45) | -20.833 (71.7433) | 31.905 (108.3337) | -25.778 (71.6205)
  Change at Week 3: SPI II (n=25, 21, 47) | -2.511 (14.1763) | 4.636 (18.1315) | -6.238 (12.4191)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 1 (Sleep disturbance): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 25.0781, 80% CI 2-sided [18.565 to 31.591], Standard Error of Mean 5.0238
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0049, Mixed Models Analysis; LS Mean Difference = 15.6481, 80% CI 2-sided [8.7110 to 22.585], Standard Error of Mean 5.3551
Statistical Analysis 3: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 1 (Snoring): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.3078, Mixed Models Analysis; LS Mean Difference = -3.6270, 80% CI 2-sided [-8.196 to 0.94237], Standard Error of Mean 3.5248
Statistical Analysis 4: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 3]; Test type: Superiority or Other; p = 0.0644, Mixed Models Analysis; LS Mean Difference = 7.1594, 80% CI 2-sided [2.2344 to 12.084], Standard Error of Mean 3.8022
Statistical Analysis 5: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 1 (ASoB): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.1517, Mixed Models Analysis; LS Mean Difference = 4.5601, 80% CI 2-sided [0.49198 to 8.6281], Standard Error of Mean 3.1318
Statistical Analysis 6: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 5]; Test type: Superiority or Other; p = 0.8252, Mixed Models Analysis; LS Mean Difference = -0.7384, 80% CI 2-sided [-5.056 to 3.5789], Standard Error of Mean 3.3281
Statistical Analysis 7: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 1 (Sleep quantity): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0063, Mixed Models Analysis; LS Mean Difference = -0.6228, 80% CI 2-sided [-0.9082 to -0.3375], Standard Error of Mean 0.2203
Statistical Analysis 8: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.3217, Mixed Models Analysis; LS Mean Difference = -0.2301, 80% CI 2-sided [-0.5283 to 0.06822], Standard Error of Mean 0.2303
Statistical Analysis 9: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 1 (Optimal sleep): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.2307, Mixed Models Analysis; LS Mean Difference = 0.1291, 80% CI 2-sided [-0.0091 to 0.26716], Standard Error of Mean 0.1065
Statistical Analysis 10: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 9]; Test type: Superiority or Other; p = 0.4585, Mixed Models Analysis; LS Mean Difference = 0.08114, 80% CI 2-sided [-0.0598 to 0.22209], Standard Error of Mean 0.1087
Statistical Analysis 11: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 1 (Sleep adequacy): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.3477, Mixed Models Analysis; LS Mean Difference = -3.6629, 80% CI 2-sided [-8.681 to 1.3549], Standard Error of Mean 3.8642
Statistical Analysis 12: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 11]; Test type: Superiority or Other; p = 0.1565, Mixed Models Analysis; LS Mean Difference = -5.8688, 80% CI 2-sided [-11.17 to -0.5693], Standard Error of Mean 4.0842
Statistical Analysis 13: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 1 (Somnolence): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.1088, Mixed Models Analysis; LS Mean Difference = -6.4319, 80% CI 2-sided [-11.55 to -1.311], Standard Error of Mean 3.9541
Statistical Analysis 14: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.8627, Mixed Models Analysis; LS Mean Difference = 0.7208, 80% CI 2-sided [-4.654 to 6.0952], Standard Error of Mean 4.1517
Statistical Analysis 15: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 1 (SPI I): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0024, Mixed Models Analysis; LS Mean Difference = 56.6310, 80% CI 2-sided [33.532 to 79.730], Standard Error of Mean 17.8056
Statistical Analysis 16: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 15]; Test type: Superiority or Other; p = 0.0112, Mixed Models Analysis; LS Mean Difference = 49.1543, 80% CI 2-sided [24.831 to 73.478], Standard Error of Mean 18.7622
Statistical Analysis 17: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 1 (SPI II): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; LS Mean Difference = 10.9197, 80% CI 2-sided [6.9105 to 14.929], Standard Error of Mean 3.0912
Statistical Analysis 18: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 17]; Test type: Superiority or Other; p = 0.0129, Mixed Models Analysis; LS Mean Difference = 8.4691, 80% CI 2-sided [4.1876 to 12.751], Standard Error of Mean 3.3037
Statistical Analysis 19: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 2 (Sleep disturbance): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis; LS Mean Difference = 14.1078, 80% CI 2-sided [8.4492 to 19.766], Standard Error of Mean 4.3667
Statistical Analysis 20: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0026, Mixed Models Analysis; LS Mean Difference = 14.3485, 80% CI 2-sided [8.4275 to 20.270], Standard Error of Mean 4.5692
Statistical Analysis 21: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 2 (Snoring): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.9305, Mixed Models Analysis; LS Mean Difference = -0.2989, 80% CI 2-sided [-4.729 to 4.1309], Standard Error of Mean 3.4103
Statistical Analysis 22: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 21]; Test type: Superiority or Other; p = 0.1178, Mixed Models Analysis; LS Mean Difference = -5.7062, 80% CI 2-sided [-10.36 to -1.050], Standard Error of Mean 3.5839
Statistical Analysis 23: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 2 (ASoB): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.3339, Mixed Models Analysis; LS Mean Difference = 2.4586, 80% CI 2-sided [-0.8124 to 5.7295], Standard Error of Mean 2.5231
Statistical Analysis 24: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 23]; Test type: Superiority or Other; p = 0.0698, Mixed Models Analysis; LS Mean Difference = 4.8590, 80% CI 2-sided [1.4493 to 8.2686], Standard Error of Mean 2.6300
Statistical Analysis 25: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 2 (Sleep quantity): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0762, Mixed Models Analysis; LS Mean Difference = -0.3364, 80% CI 2-sided [-0.5777 to -0.0950], Standard Error of Mean 0.1859
Statistical Analysis 26: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 25]; Test type: Superiority or Other; p = 0.4096, Mixed Models Analysis; LS Mean Difference = -0.1591, 80% CI 2-sided [-0.4075 to 0.08935], Standard Error of Mean 0.1913
Statistical Analysis 27: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 2 (Optimal sleep): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0455, Mixed Models Analysis; LS Mean Difference = 0.2115, 80% CI 2-sided [0.07751 to 0.34550], Standard Error of Mean 0.1033
Statistical Analysis 28: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 27]; Test type: Superiority or Other; p = 0.4585, Mixed Models Analysis; LS Mean Difference = 0.08114, 80% CI 2-sided [-0.0598 to 0.22209], Standard Error of Mean 0.1087
Statistical Analysis 29: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 2 (Sleep adequacy): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.9078, Mixed Models Analysis; LS Mean Difference = 0.5433, 80% CI 2-sided [-5.513 to 6.5995], Standard Error of Mean 4.6662
Statistical Analysis 30: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 29]; Test type: Superiority or Other; p = 0.6502, Mixed Models Analysis; LS Mean Difference = -2.1848, 80% CI 2-sided [-8.403 to 4.0338], Standard Error of Mean 4.7892
Statistical Analysis 31: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 2 (Somnolence): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.8090, Mixed Models Analysis; LS Mean Difference = -0.9029, 80% CI 2-sided [-5.716 to 3.9101], Standard Error of Mean 3.7234
Statistical Analysis 32: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 31]; Test type: Superiority or Other; p = 0.5282, Mixed Models Analysis; LS Mean Difference = 2.4351, 80% CI 2-sided [-2.532 to 7.4025], Standard Error of Mean 3.8429
Statistical Analysis 33: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 2 (SPI I): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.1848, Mixed Models Analysis; LS Mean Difference = 25.3231, 80% CI 2-sided [0.86393 to 49.782], Standard Error of Mean 18.8604
Statistical Analysis 34: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 33]; Test type: Superiority or Other; p = 0.0124, Mixed Models Analysis; LS Mean Difference = 50.4054, 80% CI 2-sided [25.134 to 75.677], Standard Error of Mean 19.4810
Statistical Analysis 35: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 2 (SPI II): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0267, Mixed Models Analysis; LS Mean Difference = 6.8658, 80% CI 2-sided [2.9504 to 10.781], Standard Error of Mean 3.0205
Statistical Analysis 36: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 35]; Test type: Superiority or Other; p = 0.0134, Mixed Models Analysis; LS Mean Difference = 8.0855, 80% CI 2-sided [3.9787 to 12.192], Standard Error of Mean 3.1677
Statistical Analysis 37: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Sleep disturbance): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0152, Mixed Models Analysis; LS Mean Difference = 9.5242, 80% CI 2-sided [4.5949 to 14.453], Standard Error of Mean 3.7993
Statistical Analysis 38: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 37]; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; LS Mean Difference = 19.9806, 80% CI 2-sided [14.602 to 25.359], Standard Error of Mean 4.1501
Statistical Analysis 39: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Snoring): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.3516, Mixed Models Analysis; LS Mean Difference = -2.7667, 80% CI 2-sided [-6.590 to 1.0562], Standard Error of Mean 2.9402
Statistical Analysis 40: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 39]; Test type: Superiority or Other; p = 0.3448, Mixed Models Analysis; LS Mean Difference = 3.0838, 80% CI 2-sided [-1.116 to 7.2838], Standard Error of Mean 3.2323
Statistical Analysis 41: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (ASoB): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.5583, Mixed Models Analysis; LS Mean Difference = -2.5882, 80% CI 2-sided [-8.294 to 3.1175], Standard Error of Mean 4.3902
Statistical Analysis 42: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 41]; Test type: Superiority or Other; p = 0.1141, Mixed Models Analysis; LS Mean Difference = 7.6547, 80% CI 2-sided [1.4717 to 13.838], Standard Error of Mean 4.7652
Statistical Analysis 43: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Sleep quantity): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0034, Mixed Models Analysis; LS Mean Difference = -0.5882, 80% CI 2-sided [-0.8356 to -0.3408], Standard Error of Mean 0.1903
Statistical Analysis 44: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 43]; Test type: Superiority or Other; p = 0.4083, Mixed Models Analysis; LS Mean Difference = -0.1722, 80% CI 2-sided [-0.4403 to 0.09599], Standard Error of Mean 0.2064
Statistical Analysis 45: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Optimal sleep): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0120, Mixed Models Analysis; LS Mean Difference = 0.2744, 80% CI 2-sided [0.13746 to 0.41127], Standard Error of Mean 0.1055
Statistical Analysis 46: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 45]; Test type: Superiority or Other; p = 0.3750, Mixed Models Analysis; LS Mean Difference = 0.1016, 80% CI 2-sided [-0.0457 to 0.24881], Standard Error of Mean 0.1136
Statistical Analysis 47: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Sleep adequacy): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.9119, Mixed Models Analysis; LS Mean Difference = 0.4367, 80% CI 2-sided [-4.665 to 5.5387], Standard Error of Mean 3.9301
Statistical Analysis 48: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 47]; Test type: Superiority or Other; p = 0.1367, Mixed Models Analysis; LS Mean Difference = -6.3429, 80% CI 2-sided [-11.79 to -0.8960], Standard Error of Mean 4.1977
Statistical Analysis 49: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (Somnolence): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.0595, Mixed Models Analysis; LS Mean Difference = -6.0062, 80% CI 2-sided [-10.05 to -1.964], Standard Error of Mean 3.1094
Statistical Analysis 50: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 49]; Test type: Superiority or Other; p = 0.1356, Mixed Models Analysis; LS Mean Difference = 5.0362, 80% CI 2-sided [0.72505 to 9.3473], Standard Error of Mean 3.3182
Statistical Analysis 51: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (SPI I): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.7528, Mixed Models Analysis; LS Mean Difference = 5.1569, 80% CI 2-sided [-15.99 to 26.303], Standard Error of Mean 16.2884
Statistical Analysis 52: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 51]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; LS Mean Difference = 67.7022, 80% CI 2-sided [45.114 to 90.290], Standard Error of Mean 17.4066
Statistical Analysis 53: Comparison: PF-03654746 (Low Dose) vs Placebo; Week 3 (SPI II): Mixed effects linear model was used with treatment, period and investigator as fixed effects; baseline as covariate and participants as random effect; Test type: Superiority or Other; p = 0.2837, Mixed Models Analysis; LS Mean Difference = 2.8582, 80% CI 2-sided [-0.5670 to 6.2835], Standard Error of Mean 2.6389
Statistical Analysis 54: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 14, analysis 53]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 12.9251, 80% CI 2-sided [9.1761 to 16.674], Standard Error of Mean 2.8913

15. Other Pre Specified Outcome: Change From Baseline in Subjective Sleep Questionnaire (SSQ) Latency Subscale Scores at Week 1, 2 and 3
Description: SSQ is a 5-item self-report scale that was designed to evaluate the amount and quality of sleep and is comprised of 5 items yielding 5 subscale scores: latency (1 item), hours of sleep (1 item), number of awakenings (1 item), total awake after sleep onset (WASO [1 item]), quality of sleep (1 item). Latency subscale score ranges from 0-840 minutes. Lower value indicates better sleep.
Time Frame: Baseline, Week 1, 2, 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 27 | 22 | 52
minutes
  Baseline (n=27, 22, 52) | 30.333 (35.7464) | 31.364 (29.7582) | 29.067 (31.8087)
  Change at Week 1 (n=25, 22, 43) | 24.6 (89.6858) | -3.409 (46.2302) | 0.837 (60.9442)
  Change at Week 2 (n=21, 19, 43) | -3.024 (23.4763) | -12.632 (31.1858) | -11.105 (23.2396)
  Change at Week 3 (n=18, 11, 36) | -3.222 (36.2086) | 4.091 (66.954) | -11.958 (30.2856)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 26.8615, 80% CI 2-sided [21.777 to 31.946], Standard Error of Mean 3.9167
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3034, Mixed Models Analysis; LS Mean Difference = 4.3455, 80% CI 2-sided [-1.080 to 9.7713], Standard Error of Mean 4.1817
Statistical Analysis 3: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0223, Mixed Models Analysis; LS Mean Difference = 6.9558, 80% CI 2-sided [3.1320 to 10.780], Standard Error of Mean 2.9408
Statistical Analysis 4: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.2284, Mixed Models Analysis; LS Mean Difference = 3.7518, 80% CI 2-sided [-0.2442 to 7.7479], Standard Error of Mean 3.0743
Statistical Analysis 5: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0201, Mixed Models Analysis; LS Mean Difference = 8.5752, 80% CI 2-sided [3.9265 to 13.224], Standard Error of Mean 3.5848
Statistical Analysis 6: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.1931, Mixed Models Analysis; LS Mean Difference = 5.0229, 80% CI 2-sided [0.07753 to 9.9683], Standard Error of Mean 3.8154

16. Other Pre Specified Outcome: Change From Baseline in Subjective Sleep Questionnaire (SSQ) Hours of Sleep Subscale Scores at Week 1, 2 and 3
Description: SSQ is a 5-item self-report scale that was designed to evaluate the amount and quality of sleep and is comprised of 5 items yielding 5 subscale scores: latency (1 item), hours of sleep (1 item), number of awakenings (1 item), WASO (1 item), quality of sleep (1 item).
  Hours of sleep subscale score ranges from 0-16 hours. Higher value indicates better sleep.
Time Frame: Baseline, Week 1, 2, 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 27 | 22 | 52
hours
  Baseline (n=27, 22, 52) | 6.05 (1.0963) | 6.48 (1.2806) | 6.364 (1.2534)
  Change at Week 1 (n=25, 22, 43) | 0.147 (1.4865) | 0.414 (2.0816) | 0.763 (1.5914)
  Change at Week 2 (21, 19, 43) | 0.414 (1.2911) | 0.319 (1.7) | 0.865 (1.4959)
  Change at Week 3 (n=18, 11, 36) | -0.148 (1.7562) | -0.17 (2.0091) | 0.717 (1.2305)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; LS Mean Difference = -0.6766, 80% CI 2-sided [-0.9046 to -0.4487], Standard Error of Mean 0.1759
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1055, Mixed Models Analysis; LS Mean Difference = -0.3075, 80% CI 2-sided [-0.5499 to -0.0650], Standard Error of Mean 0.1871
Statistical Analysis 3: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0119, Mixed Models Analysis; LS Mean Difference = -0.4684, 80% CI 2-sided [-0.7012 to -0.2356], Standard Error of Mean 0.1791
Statistical Analysis 4: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.5016, Mixed Models Analysis; LS Mean Difference = -0.1263, 80% CI 2-sided [-0.3687 to 0.11608], Standard Error of Mean 0.1866
Statistical Analysis 5: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0531, Mixed Models Analysis; LS Mean Difference = -0.3451, 80% CI 2-sided [-0.5711 to -0.1191], Standard Error of Mean 0.1738
Statistical Analysis 6: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0306, Mixed Models Analysis; LS Mean Difference = -0.4137, 80% CI 2-sided [-0.6549 to -0.1725], Standard Error of Mean 0.1856

17. Other Pre Specified Outcome: Change From Baseline in Subjective Sleep Questionnaire (SSQ) Number of Awakenings Subscale Scores at Week 1, 2 and 3
Description: SSQ is a 5-item self-report scale that was designed to evaluate the amount and quality of sleep and is comprised of 5 items yielding 5 subscale scores: latency (1 item), hours of sleep (1 item), number of awakenings (1 item), WASO (1 item), quality of sleep (1 item).
  Number of awakenings subscale score ranges from 0 to 30. Lower value indicates better sleep.
Time Frame: Baseline, Week 1, 2, 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 27 | 22 | 52
awakenings
  Baseline (n=27, 22, 52) | 1.37 (1.4317) | 1.182 (1.0065) | 1.298 (1.2258)
  Change at Week 1 (n=25, 22, 43) | 0.12 (1.6788) | 0.5 (1.7252) | -0.209 (1.4402)
  Change at Week 2 (n=21, 19, 43) | -0.333 (1.977) | 0.158 (1.2589) | -0.419 (1.2293)
  Change at Week 3 (n=18, 11, 36) | 0.028 (2.0398) | 0.045 (1.4222) | -0.361 (1.2627)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 0.7671, 80% CI 2-sided [0.54260 to 0.99157], Standard Error of Mean 0.1731
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0059, Mixed Models Analysis; LS Mean Difference = 0.5285, 80% CI 2-sided [0.28911 to 0.76798], Standard Error of Mean 0.1847
Statistical Analysis 3: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.2921, Mixed Models Analysis; LS Mean Difference = 0.1526, 80% CI 2-sided [-0.0336 to 0.33878], Standard Error of Mean 0.1431
Statistical Analysis 4: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.1929, Mixed Models Analysis; LS Mean Difference = 0.1980, 80% CI 2-sided [0.00319 to 0.39272], Standard Error of Mean 0.1498
Statistical Analysis 5: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0332, Mixed Models Analysis; LS Mean Difference = 0.3433, 80% CI 2-sided [0.13988 to 0.54663], Standard Error of Mean 0.1565
Statistical Analysis 6: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0162, Mixed Models Analysis; LS Mean Difference = 0.4184, 80% CI 2-sided [0.20006 to 0.63674], Standard Error of Mean 0.1681

18. Other Pre Specified Outcome: Change From Baseline in Subjective Sleep Questionnaire (SSQ) Total Awake After Sleep Onset (WASO) Subscale Scores at Week 1, 2 and 3
Description: SSQ is a 5-item self-report scale that was designed to evaluate the amount and quality of sleep and is comprised of 5 items yielding 5 subscale scores: latency (1 item), hours of sleep (1 item), number of awakenings (1 item), WASO (1 item), quality of sleep (1 item).
  Total WASO subscale score ranges from 0 to 24 hours. Lower value indicates better sleep.
Time Frame: Baseline, Week 1, 2, 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 27 | 22 | 52
hours
  Baseline (n=27, 22, 52) | 0.432 (0.6295) | 0.578 (0.8214) | 0.529 (0.7442)
  Change at Week 1 (25, 22, 43) | 0.109 (0.5542) | 0.013 (1.2797) | -0.286 (0.7444)
  Change at Week 2 (n=21, 19, 43) | -0.133 (0.7064) | -0.167 (0.8035) | -0.228 (0.8409)
  Change at Week 3 (n=18, 11, 36) | 0.091 (0.6291) | 0.329 (1.3329) | -0.313 (0.6863)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 0.5103, 80% CI 2-sided [0.36707 to 0.65345], Standard Error of Mean 0.1103
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0031, Mixed Models Analysis; LS Mean Difference = 0.3643, 80% CI 2-sided [0.21189 to 0.51664], Standard Error of Mean 0.1174
Statistical Analysis 3: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.1553, Mixed Models Analysis; LS Mean Difference = 0.1362, 80% CI 2-sided [0.01366 to 0.25882], Standard Error of Mean 0.09408
Statistical Analysis 4: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.2809, Mixed Models Analysis; LS Mean Difference = 0.1070, 80% CI 2-sided [-0.0205 to 0.23458], Standard Error of Mean 0.09797
Statistical Analysis 5: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0603, Mixed Models Analysis; LS Mean Difference = 0.2195, 80% CI 2-sided [0.07101 to 0.36803], Standard Error of Mean 0.1146
Statistical Analysis 6: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; LS Mean Difference = 0.4278, 80% CI 2-sided [0.27079 to 0.58479], Standard Error of Mean 0.1212

19. Other Pre Specified Outcome: Change From Baseline in Subjective Sleep Questionnaire (SSQ) Quality of Sleep Subscale Scores at Week 1, 2 and 3
Description: SSQ is a 5-item self-report scale that was designed to evaluate the amount and quality of sleep and is comprised of 5 items yielding 5 subscale scores: latency (1 item), hours of sleep (1 item), number of awakenings (1 item), WASO (1 item), quality of sleep (1 item).
  Quality of sleep subscale score ranges from 0-100. Higher score indicates better quality of sleep.
Time Frame: Baseline, Week 1, 2, 3
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 27 | 22 | 52
units on a scale
  Baseline (n=27, 22, 52) | 57.093 (19.7582) | 55 (23.4663) | 56.202 (20.9533)
  Change at Week 1 (n=25, 22, 42) | -4.06 (21.0616) | 0.5 (25.6715) | 8.393 (25.5447)
  Change at Week 2 (n=21, 19, 43) | 8.286 (22.3375) | 11.105 (22.6124) | 9.43 (20.5434)
  Change at Week 3 (n=18, 11, 36) | 7.222 (21.7764) | 0.182 (44.302) | 10.389 (22.8602)
Statistical Analysis 1: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -13.3264, 80% CI 2-sided [-16.83 to -9.828], Standard Error of Mean 2.6944
Statistical Analysis 2: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0068, Mixed Models Analysis; LS Mean Difference = -8.1260, 80% CI 2-sided [-11.87 to -4.382], Standard Error of Mean 2.8841
Statistical Analysis 3: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.1346, Mixed Models Analysis; LS Mean Difference = -3.5341, 80% CI 2-sided [-6.551 to -0.5175], Standard Error of Mean 2.3172
Statistical Analysis 4: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.6552, Mixed Models Analysis; LS Mean Difference = 1.0911, 80% CI 2-sided [-2.067 to 4.2494], Standard Error of Mean 2.4268
Statistical Analysis 5: Comparison: PF-03654746 (Low Dose) vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0765, Mixed Models Analysis; LS Mean Difference = -3.2001, 80% CI 2-sided [-5.494 to -0.9063], Standard Error of Mean 1.7614
Statistical Analysis 6: Comparison: PF-03654746 (Flexible Dose) vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0473, Mixed Models Analysis; LS Mean Difference = -3.8781, 80% CI 2-sided [-6.349 to -1.407], Standard Error of Mean 1.8976

20. Other Pre Specified Outcome: Number of Participants With Clinically Significant Laboratory Test Abnormalities
Description: Laboratory parameters included hematology (hemoglobin, hematocrit, red blood cell count, platelets, leukocytes, total neutrophils, eosinophils, basophils, lymphocytes, monocytes); liver function (total bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, albumin, total protein); renal function (creatinine, blood urea nitrogen, uric acid, sodium, potassium, chloride, bicarbonate, calcium); urinalysis (protein, blood), and clinical chemistry (glucose).
Time Frame: Baseline up to 1 week after last study dose
Population: Safety analysis set consisted of all participants who took at least 1 dose of study medication. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 28 | 25 | 55
participants | 5 | 9 | 10

21. Other Pre Specified Outcome: Number of Participants With Electrocardiogram (ECG) Findings
Description: Criteria for potential clinical concern in ECG parameters: maximum PR interval of greater than or equal to (>=) 300 milliseconds (msec), maximum QRS interval >=200 msec, maximum QTc interval of 450 to <480 msec, 480 to <500 msec and >=500 msec.
Time Frame: Baseline up to End of Treatment (Week 3 of period 2)
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 28 | 25 | 57
participants | 1 | 0 | 1

22. Other Pre Specified Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities
Description: Criteria for potential clinical concern in vital signs: systolic blood pressure (BP) less than (<) 90 millimeters of mercury (mmHg), diastolic BP <50 mmHg, supine and sitting heart rate <40 beats per minute (bpm) or >120 bpm, standing and erect heart rate <40 bpm or >140 bpm. Maximum increase from baseline in systolic BP >=30 mmHg, maximum increase from baseline in diastolic BP >=20 mmHg.
Time Frame: Baseline up to 1 week after last study dose
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 28 | 25 | 55
participants | 0 | 0 | 1

23. Other Pre Specified Outcome: Number of Participants With Change From Baseline in Physical Examination and Neurological Examination
Description: Analysis include general physical examination and assessment of head, ears, eyes, ocular fundi, nose, mouth, throat, neck, thyroid, lungs, heart, breasts, abdomen and musculoskeletal system.
Time Frame: Baseline up to 1 week after last study dose (1 week after end of Period 2)
Population: Safety analysis set consisted of all participants who took at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 28 | 25 | 58
participants | 0 | 0 | 0

24. Other Pre Specified Outcome: Treatment Duration
Description: Treatment duration was defined as the total number of dosing days from first to last day of study drug administration in each period.
Time Frame: Day 1 up to Day 21
Population: Safety analysis set consisted of all participants who took at least 1 dose of study medication.
Measure: Mean (Full Range); unit: days
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Number analyzed (Participants) | 28 | 25 | 58
days | 21 [1 to 30] | 21 [7 to 27] | 21 [3 to 45]

ADVERSE EVENTS:
Description: Safety analysis population included all participants who received at least 1 dose of study medication.
Arm/Group | PF-03654746 (Low Dose) | PF-03654746 (Flexible Dose) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/25 | 0/58
Other Adverse Events (participants affected / at risk) | 21/28 | 19/25 | 33/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03654746 (Low Dose) (N=28) | PF-03654746 (Flexible Dose) (N=25) | Placebo (N=58)
Palpitations (Cardiac disorders) | 1 | 1 | 0
Hyperacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 2
Fatigue (General disorders) | 1 | 1 | 10
Feeling abnormal (General disorders) | 0 | 0 | 2
Feeling jittery (General disorders) | 1 | 0 | 0
Irritability (General disorders) | 2 | 2 | 3
Pyrexia (General disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood albumin increased (Investigations) | 0 | 1 | 0
Blood amylase increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Coordination abnormal (Nervous system disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 2 | 10
Memory impairment (Nervous system disorders) | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 1 | 0
Poor quality sleep (Nervous system disorders) | 0 | 1 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 2 | 3 | 3
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 1
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 1
Impatience (Psychiatric disorders) | 0 | 1 | 0
Initial insomnia (Psychiatric disorders) | 2 | 2 | 3
Insomnia (Psychiatric disorders) | 9 | 4 | 4
Libido decreased (Psychiatric disorders) | 1 | 0 | 1
Middle insomnia (Psychiatric disorders) | 0 | 1 | 1
Nervousness (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
Instead of time to sustained response, data for percentage of sustained responders in time-sensitive ADHD symptom scale (TASS) total score was reported as per planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.